CLINICAL TRIAL: NCT06511674
Title: Vulnerability and Risk of Neuropathic Pain in Cancer: Validation of a Predictive Tool to Optimize Treatment.
Brief Title: Vulnerability and Risk of Neuropathic Pain in Cancer
Acronym: CANOPY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RBHP 2023 PICKERING
Record Dates: First submitted 2024-07-04; First posted 2024-07-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-06

CONDITIONS: Neuropathic Pain; Cancer; Predictive
MeSH Terms: conditions — Neuralgia; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Cancer patients and Healthy Volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer patients (Experimental): 500 cancer patients: 100 women with breast cancer, 100 women with gynecological cancer, 150 patients with lung cancer (100 men, 50 women) and 150 patients with colorectal cancer (100 men, 50 women).
  Interventions: Other: Cognitive-emotional and pain assessments
- Healthy volunteers controls (Experimental): 125 healthy control volunteers from the volunteer database
  Interventions: Other: Cognitive-emotional and pain assessments

INTERVENTIONS:
Other: Cognitive-emotional and pain assessments — Data collection on cognitive-emotional and pain parameters using questionnaires.

SUMMARY:
Successive and repeated therapeutic interventions during cancer management - surgery, chemotherapy, radiotherapy - can all, to varying degrees, generate acute pain, central pain sensitization and chronic pain. Almost 58% of patients suffer from chronic pain, often of the neuropathic type, with altered quality of life and disease burden amplified by difficulty in achieving effective relief.

Indeed, neuropathic pain in cancer remains difficult to treat, often arrives insidiously, may persist well beyond cancer remission, and frequently has a fate that is difficult to predict. Current treatments for neuropathic pain are based on the recommendations of learned societies, but therapeutic failures are frequent, and iatrogenic pathology is high. Many factors have been identified as being associated with the development of chronic pain in cancer patients. The intensity of preoperative pain, opioid consumption, age, sleep disorders, cognitive-emotional state, psychological vulnerability and social precariousness are all factors that influence and perpetuate chronic pain linked to cancer and its management. Several studies have shown that 6 months or 1 year after cancer diagnosis, there are various pain trajectories, enabling us to identify several pain patient phenotypes. The patient's overall state of vulnerability at the time of cancer diagnosis has an impact on the trajectory of pain chronicisation, and it is often difficult for clinicians to apprehend this risk. In practice, we lack a validated, easy-to-use tool that would enable us to predict the risk of pain chronicisation for each patient, even before the start of the treatment process.

ELIGIBILITY:
Inclusion Criteria Patients:

* Patient over 18 years of age,
* Patient suffering from cancer (breast, gynecological, colorectal, lung) and having to undergo one or more anti-cancer therapeutic procedures (chemotherapy, surgery, hormonal therapy, radiotherapy, targeted therapy, etc.),
* Sufficient cooperation and understanding to comply with the study requirements,
* Agreement to give oral consent for the study,
* Affiliation with the French Social Security system.

Exclusion Criteria Patients:

* History of cancer and anti-cancer therapy (surgery, chemotherapy, radiotherapy, hormone therapy, targeted therapy, etc.),
* History and/or presence of primary brain tumors (glioblastoma, meningioma, neurofibroma, etc.) ),
* History of neurological disorders (Parkinson's disease, Alzheimer's disease, dementia, epilepsy, moderate to severe head trauma, etc.),
* Medical and/or surgical history judged by the investigator or his representative to be incompatible with the study,
* Subject whose cooperation and understanding do not allow strict compliance with the conditions laid down in the protocol,
* Pregnant or breast-feeding women,
* Beneficiary of a legal protection measure.

Inclusion Criteria Healthy Volunteers:

* Subject over 18 years of age,
* Subject free of any treatment in the 7 days preceding inclusion, in particular no use of analgesics, or judged by the investigator or his representative to be compatible with the study
* Subject with no history of cancer,
* Subject considered to be in good health by the investigator,
* Sufficient cooperation and understanding to comply with the study requirements,
* Agreement to give oral consent to the study,
* Affiliation with the French Social Security system,

Exclusion Criteria Healthy Volunteers:

* Subjects with a medical and/or surgical history judged by the investigator or his representative to be incompatible with the trial,
* Subjects whose cooperation and understanding do not allow strict compliance with the conditions laid down in the protocol,
* Pregnant or breast-feeding woman,
* Participating in another clinical trial, or within the exclusion period, or having received a total amount of compensation exceeding 4500 euros over the 12 months preceding the start of the trial,
* Benefiting from a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 625 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
CANoPy score (Z-score) | Baseline
  Calculation of the CANoPy score (Z-score) predictive of the development of neuropathic pain.
  The z-scores are then averaged across endpoints for each patient.
CANoPy score (Z-score) | 6 months
  Calculation of the CANoPy score (Z-score) predictive of the development of neuropathic pain.
  The z-scores are then averaged across endpoints for each patient.
CANoPy score (Z-score) | 12 months
  Calculation of the CANoPy score (Z-score) predictive of the development of neuropathic pain.
  The z-scores are then averaged across endpoints for each patient.

SECONDARY OUTCOMES:
Pain assessment using the Numerical Pain Scale (EN) | Baseline
  Numerical Pain Scale (EN): This numerical scale provides a pain assessment from 0 to 10.
Pain assessment using the Neuropathic Pain Questionnaire (DN4) | Baseline
  Neuropathic Pain (DN4): This questionnaire estimates the probability of neuropathic pain in a patient, by means of four questions divided into ten items to be ticked. The practitioner or clinical research associate in charge of the study interviews or examines the patient and fills in the questionnaire himself. Each item is marked with a "yes" or "no" answer. Each "yes" is worth a score of 1, and each "no" is worth a score of 0. The sum of the scores gives the patient's score (out of 10); if the patient's score is equal to or greater than 4/10, the test is positive.
Pain assessment using the Numerical Pain Scale (EN) | 6 months
  Numerical Pain Scale (EN): This numerical scale provides a pain assessment from 0 to 10.
Pain assessment using the Neuropathic Pain Questionnaire (DN4) | 6 months
  Neuropathic Pain (DN4): This questionnaire estimates the probability of neuropathic pain in a patient, by means of four questions divided into ten items to be ticked. The practitioner or clinical research associate in charge of the study interviews or examines the patient and fills in the questionnaire himself. Each item is marked with a "yes" or "no" answer. Each "yes" is worth a score of 1, and each "no" is worth a score of 0. The sum of the scores gives the patient's score (out of 10); if the patient's score is equal to or greater than 4/10, the test is positive.
Pain assessment using the Numerical Pain Scale (EN) | 12 months
  Numerical Pain Scale (EN): This numerical scale provides a pain assessment from 0 to 10.
Pain assessment using the Neuropathic Pain Questionnaire (DN4) | 12 months
  Neuropathic Pain (DN4): This questionnaire estimates the probability of neuropathic pain in a patient, by means of four questions divided into ten items to be ticked. The practitioner or clinical research associate in charge of the study interviews or examines the patient and fills in the questionnaire himself. Each item is marked with a "yes" or "no" answer. Each "yes" is worth a score of 1, and each "no" is worth a score of 0. The sum of the scores gives the patient's score (out of 10); if the patient's score is equal to or greater than 4/10, the test is positive.
Assessment of cognitive status using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-COG) questionnaire | Baseline
  Functional Assessment of Cancer Therapy COGnitive function (FACT-COG): The Functional Assessment of Cancer Therapy-COGnitive function, known as FACT-COG, is a 37-item self-report questionnaire of perceived cognitive impairment. It assesses mental acuity, attention and concentration, memory, verbal fluency, functional interference, deficits observed by others, changes from previous functioning and impact on quality of life. These items were developed on the basis of interviews with cancer patients and their carers. The FACT-COG has been validated in a study of cancer patients.
Assessment of cognitive status using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-COG) questionnaire | 6 months
  Functional Assessment of Cancer Therapy COGnitive function (FACT-COG): The Functional Assessment of Cancer Therapy-COGnitive function, known as FACT-COG, is a 37-item self-report questionnaire of perceived cognitive impairment. It assesses mental acuity, attention and concentration, memory, verbal fluency, functional interference, deficits observed by others, changes from previous functioning and impact on quality of life. These items were developed on the basis of interviews with cancer patients and their carers. The FACT-COG has been validated in a study of cancer patients.
Assessment of cognitive status using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-COG) questionnaire | 12 months
  Functional Assessment of Cancer Therapy COGnitive function (FACT-COG): The Functional Assessment of Cancer Therapy-COGnitive function, known as FACT-COG, is a 37-item self-report questionnaire of perceived cognitive impairment. It assesses mental acuity, attention and concentration, memory, verbal fluency, functional interference, deficits observed by others, changes from previous functioning and impact on quality of life. These items were developed on the basis of interviews with cancer patients and their carers. The FACT-COG has been validated in a study of cancer patients.
Assessment of emotional status using the Anxiety and Depression Scale (HAD) | Baseline
  The Hospital Anxiety Depression (HAD) scale is a 14-item self-administered questionnaire completed by the patient. These items are divided into two subscales: 7 items to assess depression and 7 items to assess anxiety.
Assessment of emotional status using the Anxiety and Depression Scale (HAD) | 6 months
  The Hospital Anxiety Depression (HAD) scale is a 14-item self-administered questionnaire completed by the patient. These items are divided into two subscales: 7 items to assess depression and 7 items to assess anxiety.
Assessment of emotional status using the Anxiety and Depression Scale (HAD) | 12 months
  The Hospital Anxiety Depression (HAD) scale is a 14-item self-administered questionnaire completed by the patient. These items are divided into two subscales: 7 items to assess depression and 7 items to assess anxiety.
Evaluation of social vulnerability using the questionnaire Evaluation of Deprivation and Inequalities in Health Examination Centres (EPICES) | Baseline
  The Evaluation of Deprivation and Inequalities in Health Examination Centres (EPICES) questionnaire consists of 11 binary questions (yes/no) used to calculate an individual score indicating precariousness and health inequalities ranging from 0 to 100.
Evaluation of social vulnerability using the questionnaire Evaluation of Deprivation and Inequalities in Health Examination Centres (EPICES) | 6 months
  The Evaluation of Deprivation and Inequalities in Health Examination Centres (EPICES) questionnaire consists of 11 binary questions (yes/no) used to calculate an individual score indicating precariousness and health inequalities ranging from 0 to 100.
Evaluation of social vulnerability using the questionnaire Evaluation of Deprivation and Inequalities in Health Examination Centres (EPICES) | 12 months
  The Evaluation of Deprivation and Inequalities in Health Examination Centres (EPICES) questionnaire consists of 11 binary questions (yes/no) used to calculate an individual score indicating precariousness and health inequalities ranging from 0 to 100.
Assessment of quality of life using the EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) | Baseline
  EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) : The self-reported EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) is used as a tool to measure the (health-related) quality of life of cancer patients. This tool is used to assess their own level of functioning in different areas of quality of life.The questionnaire comprises 9 subscales, each consisting of several items: 5 subscales measuring functional status, 3 symptom subscales, and an overall subscale measuring quality of life and state of health.
Assessment of quality of sleep using the Pittsburgh Sleep Quality Index (PSQI) | Baseline
  Pittsburg Sleep Quality Index (PSQI): The Pittsburg Sleep Quality Index (PSQI) is a self-administered questionnaire comprising 19 items. It was developed to measure sleep quality in the month preceding the patient interview. The questionnaire has 7 components: subjective sleep quality, sleep latency, sleep duration, usual sleep efficiency, sleep disturbance, use of sleep medication and poor daytime sleepiness.
Assessment of quality of life using the EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) | 6 months
  EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) : The self-reported EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) is used as a tool to measure the (health-related) quality of life of cancer patients. This tool is used to assess their own level of functioning in different areas of quality of life.The questionnaire comprises 9 subscales, each consisting of several items: 5 subscales measuring functional status, 3 symptom subscales, and an overall subscale measuring quality of life and state of health.
Assessment of quality of sleep using the Pittsburgh Sleep Quality Index (PSQI) | 6 months
  Pittsburg Sleep Quality Index (PSQI): The Pittsburg Sleep Quality Index (PSQI) is a self-administered questionnaire comprising 19 items. It was developed to measure sleep quality in the month preceding the patient interview. The questionnaire has 7 components: subjective sleep quality, sleep latency, sleep duration, usual sleep efficiency, sleep disturbance, use of sleep medication and poor daytime sleepiness.
Assessment of quality of life using the EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) | 12 months
  EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) : The self-reported EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) is used as a tool to measure the (health-related) quality of life of cancer patients. This tool is used to assess their own level of functioning in different areas of quality of life.The questionnaire comprises 9 subscales, each consisting of several items: 5 subscales measuring functional status, 3 symptom subscales, and an overall subscale measuring quality of life and state of health.
Assessment of quality of sleep using the Pittsburgh Sleep Quality Index (PSQI) | 12 months
  Pittsburg Sleep Quality Index (PSQI): The Pittsburg Sleep Quality Index (PSQI) is a self-administered questionnaire comprising 19 items. It was developed to measure sleep quality in the month preceding the patient interview. The questionnaire has 7 components: subjective sleep quality, sleep latency, sleep duration, usual sleep efficiency, sleep disturbance, use of sleep medication and poor daytime sleepiness.
Assessment of disease perception and beliefs using the Illness Perception Questionnaire Revised (IPQ-R) | Baseline
  Illness Perception Questionnaire Revised (IPQ-R): The Illness Perception Questionnaire Revised (IPQ-R) is a self-administered questionnaire which assesses representations of the illness. It consists of 70 items divided into three categories: vision of the illness, point of view of the illness and causes of the illness.
Assessment of disease perception and beliefs using the disease-specific Cancer Locus of Control Scale (CLCS) | Baseline
  Cancer Locus of Control Scale (CLCS): This 17-item disease-specific controllability scale has been validated in a French population of breast cancer patients and is used to measure the perception of control over serious chronic illness and cancer. The items are rated using a four-point Likert scale (from 1 "strongly disagree" to 4 "strongly agree"). The items are divided into three subscales: perceived control over the course of the disease, internal causal attribution, and religious control.
Assessment of disease perception and beliefs using the Illness Perception Questionnaire Revised (IPQ-R) | 6 months
  Illness Perception Questionnaire Revised (IPQ-R): The Illness Perception Questionnaire Revised (IPQ-R) is a self-administered questionnaire which assesses representations of the illness. It consists of 70 items divided into three categories: vision of the illness, point of view of the illness and causes of the illness.
Assessment of disease perception and beliefs using the disease-specific Cancer Locus of Control Scale (CLCS) | 6 months
  Cancer Locus of Control Scale (CLCS): This 17-item disease-specific controllability scale has been validated in a French population of breast cancer patients and is used to measure the perception of control over serious chronic illness and cancer. The items are rated using a four-point Likert scale (from 1 "strongly disagree" to 4 "strongly agree"). The items are divided into three subscales: perceived control over the course of the disease, internal causal attribution, and religious control.
Assessment of disease perception and beliefs using the Illness Perception Questionnaire Revised (IPQ-R) | 12 months
  Illness Perception Questionnaire Revised (IPQ-R): The Illness Perception Questionnaire Revised (IPQ-R) is a self-administered questionnaire which assesses representations of the illness. It consists of 70 items divided into three categories: vision of the illness, point of view of the illness and causes of the illness.
Assessment of disease perception and beliefs using the disease-specific Cancer Locus of Control Scale (CLCS) | 12 months
  Cancer Locus of Control Scale (CLCS): This 17-item disease-specific controllability scale has been validated in a French population of breast cancer patients and is used to measure the perception of control over serious chronic illness and cancer. The items are rated using a four-point Likert scale (from 1 "strongly disagree" to 4 "strongly agree"). The items are divided into three subscales: perceived control over the course of the disease, internal causal attribution, and religious control.
Assessment of analgesic consumption | Baseline
  Assessment of analgesic consumption throughout the study.
Assessment of analgesic consumption | 6 months
  Assessment of analgesic consumption throughout the study.
Assessment of analgesic consumption | 12 months
  Assessment of analgesic consumption throughout the study.

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - Centre Hospitalier d'Ajaccio, Ajaccio
  - Centre de Lutte contre le Cancer - Institut de Cancérologie de l'Ouest, Angers
  - Centre Hospitalier Henri Mondor d'Aurillac, Aurillac
  - Centre de Lutte contre le Cancer - Institut Bergonié, Bordeaux
  - Centre de Lutte contre le Cancer - Centre François Baclesse, Caen
  - Centre Hospitalier Universitaire Caen Normandie, Caen
  - Centre de Lutte contre le Cancer - Jean Perrin, Clermont-Ferrand
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpitaux civils de Colmar, Colmar
  - Centre Régional de Lutte contre le Cancer - Georges Francois Leclerc, Dijon
  - Hôpital privé le Bois, Lille
  - Centre Hospitalier de Montluçon, Montluçon
  - Centre Hospitalier de Moulins-Yzeure, Moulins
  - Hôpital Saint-Louis APHP, Paris
  - Hôpital Beaujon AP-HP, Paris
  - Institut Godinot, Reims
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - CH Valenciennes, Valenciennes
  - Institut Gustave Roussy, Villejuif